CLINICAL TRIAL: NCT02908802
Title: A Double-Blind Placebo Controlled Study of Probiotic Supplement as Treatment for Students With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Probiotic Supplement as Treatment for Students With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 40-16
Record Dates: First submitted 2016-09-18; First posted 2016-09-21 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Probiotic capsules: two capsules twice a day
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Probiotic capsules without the active ingredient: two capsules twice a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic
  Arms: Probiotic
Dietary Supplement: Placebo — Probiotics capsules without the active ingredient
  Arms: Placebo

SUMMARY:
Subjects will answer the following questionnaire and tests:

* Symptom severity and improvement will be measured using ADHA Rating scale IV (ADHD RS)
* Demographic Questionnaire - composed by the researchers
* Family Eating Habits Questionnaire (FEAHQ-33)
* Food Frequency Questionnaire (FFQ)
* Test MOXO

The subjects will take the study product for six months.

After six months the subject will fill once again all the questionnaires.

DETAILED DESCRIPTION:
Computerized performance test MOXO - the test has been developed in Israel by Neurotech Company. The test's goal is to assess and define a participant's performance according to the four indices of Attention Deficit Hyperactivity Disorder: Attention, Hyperactivity, Impulsivity, and Timing with adjustment for age.

Subjects will answer the following questionnaire and tests:

* Symptom severity and improvement will be measured using ADHA Rating scale IV (ADHD RS)
* Demographic Questionnaire - composed by the researchers
* Family Eating Habits Questionnaire (FEAHQ-33)
* Food Frequency Questionnaire (FFQ)
* Test MOXO

The subjects will take the study product for six months.

After six months the subject will fill once again all the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Students registered in the college's Support Center for Students with Learning Disabilities and who have been diagnosed by a computerized didactic assessment -MATAL - as well as an attention diagnosis by a psychiatrist or a neurologist,
* Students who are not treated by medication or alternative treatment,
* Students who are not due to complete their education at Tel Hai College during the study period,
* Students who have signed on an informed consent form,
* No dairy intolerance (student can consume milk without any adverse effects),
* No soy allergy,
* Not currently taking any antibiotics or probiotics,
* Not pregnant or planning to become pregnant during the study period,
* Not been diagnosed with any of the following:

  * Cancer
  * HIV/AIDS
  * Crohn's disease
  * Ulcerative colitis
  * Immune compromised illness
  * Other serious illness

Exclusion Criteria:

* Students treated by any type of treatment for Attention Deficit Hyperactivity Disorder,
* Students who have not been assessed by MATAL and a psychiatrist,
* Students who take antibiotics.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Reduce symptoms of attention deficit measured by MOXO test | Six month
  After six month of treatment reduce symptoms of attention deficit will be measured by MOXO test

CONTACTS AND LOCATIONS:
Overall Officials: Snait Tamir, Professor, Study Director — snait@telhai.ac.il

IPD SHARING:
Plan to Share IPD: No